CLINICAL TRIAL: NCT05014399
Title: Cognitive Impairment in Colorectal Cancer Patients Receiving Cytotoxic Chemotherapy
Acronym: Chemo Brain
Status: Recruiting | Type: Observational
Sponsor: Joseph McCollom (Other)
Collaborators: Indiana University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Joseph McCollom, Oncologist, Parkview Health
Organization: Parkview Health (Other)
Other Study IDs: PRC-ONCOLOGY-21-0628-PPG
Record Dates: First submitted 2021-08-03; First posted 2021-08-20 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Neoplasm, Colorectal; Cognitive Impairment; Cognitive Dysfunction; Cognitive Change; Chemo-brain; Chemo Fog; Chemotherapy Effect; Cognitive Decline
Keywords: Palliative Care; Palliative Oncology; Supportive Care; Supportive Oncology; Cognitive Impairment; Chemo Brain
MeSH Terms: conditions — Colorectal Neoplasms; Cognitive Dysfunction; Chemotherapy-Related Cognitive Impairment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this research study is to see how the brain changes in patients receiving chemotherapy (cytotoxic drug) treatment for colon or rectal cancer at Parkview Cancer Institute. This information will be used to identify helpful tests to diagnose individuals at risk for developing difficulties with thinking and memory due to their cancer treatments.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained and documented according to International Conference on Harmonisation (ICH)- Good Clinical Practice (GCP), the local regulatory requirements, and permission to use private health information in accordance with the Health Insurance Portability and Accountability Act (HIPAA) prior to study-specific screening procedures. Must be able to provide study-specific informed consent prior to study entry.
* A histologically-confirmed colorectal tumor
* Patients who will be treated with cytotoxic chemotherapies including Capecitabine, Oxaliplatin, 5 fluorouracil, and Irinotecan are eligible.
* Patients must not have received cytotoxic chemotherapy previous to enrollment.

Exclusion Criteria:

* Prior administration of anti-cancer chemotherapy, radiotherapy, immunotherapy, or investigational agents
* Patients having mental incompetence as assessed by study PI, which would hinder completion of the surveys
* Pregnant or breastfeeding
* Any known brain metastases
* Non-English speaking patients
* Patients who have been diagnosed with any neuro-cognitive disorder including traumatic brain injuries, Alzheimer's disease, Parkinson's disease, Huntington's disease, and Creutzfeldt-Jakob disease.
* Patients deemed inappropriate to participate in this study by the study PI or coordinator will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All self representation of gender identity accepted
Study Population: Ambulatory colorectal oncology patients undergoing cytotoxic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Survey | 7 Years
  FACT-Cog V3
The Proteome Profiler Human XL Cytokine Array Kit (https://www.rndsystems.com/products/proteome-profiler-human-xl-cytokine-array-kit_ary022b) | 7 years
  This panel of plasma factors will be will be used to detect protein from the blood of patients throughout and after chemotherapy treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McCollom, DO, Principal Investigator — Parkview Health
Locations (1):
- Parkview Cancer Institute, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No